CLINICAL TRIAL: NCT06500741
Title: Discrete Choice Experiment to Assess the Preferences for Novel Hormonal Therapy and Androgen-deprivation Therapy in Patients With Prostate Cancer
Brief Title: Experiment to Assess Preferences for Novel Hormonal Therapy and Androgen-deprivation Therapy in Prostate Cancer Patients
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 9785-MA-3547
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Novel hormonal therapy; Androgen-deprivation therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Participants will include urologists or oncologists for the physician interviews and prostate cancer patients for the patient interviews and surveys.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No investigational drug will be administered to participants in this study.

SUMMARY:
The purpose of this study is to quantify the preferences for novel hormonal therapy (NHT) +/- androgen-deprivation therapy (ADT) vs ADT monotherapy among patients with non-metastatic hormone-sensitive prostate cancer (PC) in the United States (US), Germany, Spain, France, Italy, the United Kingdom (UK), South Korea, Australia, and Brazil, using a discrete choice experiment (DCE).

DETAILED DESCRIPTION:
The study will collect data from eligible patients (six total) and physicians (six total) from one-on-one qualitative interviews and eligible patients from online surveys. Approximately 330 patients with PC will be recruited to complete the online DCE survey.

ELIGIBILITY:
Inclusion Criteria:

Physician inclusion criteria

* The physician is a certified urologist or oncologist. The final selection will be adjusted to local practice.
* The physician has cared for at least ten nmHSPC patients in the past year.
* The physician has experience prescribing NHT and ADT. Patient inclusion criteria
* The patient has nmHSPC after radiotheraphy (RT) and/or radical prostatectomy (RP), defined as an adult patient with nmPC who had RT and/or RP.

Exclusion Criteria:

Physician exclusion criteria

* None Patient exclusion criteria
* The patient is castration resistant.
* The patient has metastatic PC.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult prostate cancer patients and urologists or oncologists who have cared for at least ten non-metastatic hormone-sensitive prostate cancer (nmHSPC) patients in the past year.
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Patients' Preference weights for different treatment attributes | Up to 1 day
  Preference data will be collected via online survey questionnaires designed using DCE method.
Patients' Overall Preference for a specific treatment profile (NHT +/- ADT or ADT monotherapy) | Up to 1 day
  Preference data will be collected via online survey questionnaires designed using DCE method.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Analysis Group, Inc., Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.